CLINICAL TRIAL: NCT01417377
Title: Non-Interventional Study to Document the Efficacy in Routine Clinical Practice of Mircera in Pakistan (NORM)
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-epoetin Beta) in Anemic Patients With Chronic Kidney Disease (NORM)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25368
Record Dates: First submitted 2011-08-05; First posted 2011-08-16 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort: Mircera
  Interventions: Drug: Mircera

INTERVENTIONS:
Drug: Mircera — Participants with chronic kidney disease receiving methoxy polyethylene glycol-epoetin beta (Mircera) and previously on treatment with short-acting epoetin alpha will be observed for a period of 6 months.

SUMMARY:
This observational, prospective, multi-centre, single-arm study will evaluate the efficacy of Mircera (methoxy polyethylene glycol-epoetin beta) in patients with chronic kidney disease previously on treatment with short-acting epoetin alpha. Data will be collected for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 18 years or above
* Chronic kidney disease (CKD) with anemia
* Patients on dialysis receiving short-acting epoetin (EPO)
* Serum ferritin level >/=100 ng/ml or transferrin saturation (TSAT) >/=20%

Exclusion Criteria:

* Patients unwilling to give informed consent
* Uncontrolled hypertension
* Transfusion of red blood cells within 8 weeks of the start of Mircera treatment
* Relevant acute or chronic bleeding history
* Hemolysis
* Hemoglobinopathies
* Pure red cell aplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Pakistan (6):
  - Sheikh Zayed Hospital; Department of Nephrology, Lahore
  - Fatima Memorial Hospital; Nephrology, Lahore
  - Doctor's Hospital and Medical Centre, Lahore
  - Khair-un-Nisa Hospital, Lahore
  - Surgimed Hospital, Lahore
  - Northwest General Hospital; Department of Nephrology, Peshawar

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera: Participants with chronic kidney disease receiving methoxy polyethylene glycol-epoetin beta (Mircera) and previously on treatment with short-acting epoetin alpha were observed for a period of 6 months.
Period: Overall Study
Arm/Group | Mircera
Started | 22
Treated | 21
Completed | 9
Not Completed | 13
Not completed — Lost to Follow-up | 12
Not completed — Enrolled, but not treated | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who were enrolled in the study. Age (continuous) data were reported only for treated participants.
Arm/Group | Mircera
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of participants analyzed for this baseline characteristic were 21, as the age data were available only for treated participants.
  years | 55.2 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Hemoglobin (Hb) Levels Between 11-12 Gram Per Deciliter (g/dL) During Final 2 Months of Study
Time Frame: Month 4 up to Month 6
Population: None of the enrolled participants in the study achieved Hb level between 11 to 12 g/dL during the final 2 months of study, therefore this particular endpoint was not analyzed.
Arm/Group | Mircera
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Achieve Hb Level to 11-12 g/dL
Time Frame: Up to 6 months
Population: as for outcome 1
Arm/Group | Mircera
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Dose Adjustments Required to Maintain Hb Levels
Time Frame: Up to 6 months
Population: as for outcome 1
Arm/Group | Mircera
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Doses of Mircera Taken as Per the Schedule in Summary of Product Characteristics (SmPC)
Time Frame: Up to 6 months
Population: The number of doses were not collected because the participants never achieved Hb level of 11 to 12 g/dL.
Arm/Group | Mircera
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Mircera
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=22)
Cardio-respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=22)
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Gastroenteritis (Gastrointestinal disorders) | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
As none of the enrolled participants in the study achieved the endpoint of maintaining Hb level between 11-12 g/dL during the final 2 months of study, therefore efficacy parameters were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.